CLINICAL TRIAL: NCT05703893
Title: Investigation of the Neurovegetative Pattern in the Adult Population With Thoracic Aortic Aneurysms (AAT)
Brief Title: Investigation of the Neurovegetative Pattern in Patients With Thoracic Aortic Aneurysms (TAA)
Acronym: IPaNeMA
Status: Active, not recruiting | Type: Observational
Sponsor: IRCCS Policlinico S. Donato (Other)
Collaborators: Politecnico di Milano (Other)
Responsible Party: Principal Investigator, Alessandro Pini, Principal Investigator, IRCCS Policlinico S. Donato
Other Study IDs: IPaNeMA
Record Dates: First submitted 2023-01-10; First posted 2023-01-30 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Rare Diseases; Aortic Aneurysm, Thoracic
Keywords: Thoracic Aneurysms; Heart rate Variability; Autonomic Nervous System
MeSH Terms: conditions — Rare Diseases; Aortic Aneurysm, Thoracic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Syndromic TAA: Patients presenting either clinical or genetic phenotype referring to a syndrome related to Thoracic Aortic Aneurysms
  Interventions: Diagnostic Test: Supine resting (REST) and active standing (STAND)
- Non-syndromic TAA: Patients presenting Thoracic Aortic Aneurysms
  Interventions: Diagnostic Test: Supine resting (REST) and active standing (STAND)

INTERVENTIONS:
Diagnostic Test: Supine resting (REST) and active standing (STAND) — Analysis of baroreflex sensitivity

SUMMARY:
The goal of this observational cross-sectional study is to learn about vagal features in patients with syndromic and non-syndromic TAA. The main question it aims to answer is to highlight a functional condition that could help stratify patients with TAA on the risk of aortic complications.

Participant will take part by standing in supine position for 10 minutes and during active standing for 10 minutes. In this period of time, it will be possible to acquire the signals continuously and non invasively through recorded non-invasive blood pressure and piezoelectric sensor breathing belt.

DETAILED DESCRIPTION:
Changes in blood pressure (BP) are tightly controlled by a neural surveillance system that triggers changes in response to heart rate, vascular tone, and respiration.

Therefore, studies in literature have investigated the regulatory effects of the sympathetic system on the tone of the vessels as well as on the BP, but further analysis are needed in order to describe its potential impact on the structure of the aortic wall and, in particular, its potential implications on aneurysms and risk of aortic dissections.

Considering that, in the population with TAA, the neurovegetative pattern influences the responses to different stressors (environmental, occupational and emotional) and also acts on the BP, which represents a risk factor for the TAA population, its analysis would allow to identify attitudes and behavioral predispositions and therefore response to stressors.

The non-invasive analysis of sympatho-adrenergic patterns could help to highlight a functional condition related to the "environmental stressors" which could help to stratify patients with TAA based on the level of pathological reactivity with effects on risk of aortic complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65 years with syndromic and nonsyndromic TAA;
* Signed informed consent;
* Patients on regular pharmacological prophylaxis (with Losartan) or naïve patients with a first diagnosis

Exclusion Criteria:

* Acute and chronic inflammatory diseases such as: liver disease, chronic renal insufficiency (creatinine > 1.5 mg/dl) and diseases affecting the thyroid system.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary care clinic, hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 139 (Estimated)
Dates: Start 2021-11-09 (Actual); Primary Completion 2024-10-25 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Supine resting (REST) and active standing (STAND) | 18 months
  Baroreflex sensitivity

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Policlinico San Donato, San Donato Milanese, Lombardy, Italy